CLINICAL TRIAL: NCT05422846
Title: Investigation of the Effect of Different Exercise Training on Wound Healing ın Patients With Diabetic Foot Ulcer
Brief Title: Investigation of the Effects of Different Exercise on Wound Healing in Patients wıth Diabetic Foot Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harran University (Other)
Responsible Party: Principal Investigator, Fatih Enzin, Principal Investigator, Harran University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: diabetic rehabilitation
Record Dates: First submitted 2022-06-06; First posted 2022-06-21 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Diabetic Foot Ulcer; Wound
Keywords: diabetes mellitus, exercise, ulcer
MeSH Terms: conditions — Diabetic Foot; Wounds and Injuries; Diabetes Mellitus; Motor Activity; Ulcer | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Two groups to be applied two different exercises progressing together with the control group
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- exercise protocol group (Experimental): The group that applied progressive exercise according to the motivation of patients and healing status of ulcers.
  Interventions: Other: exercise protocol
- aerobic exercise group (Experimental): The group performing aerobic exercise with a bicycle ergometer
  Interventions: Other: aerobic exercise
- control group (Experimental): The group to which standard applications of DFU treatment will be applied
  Interventions: Other: standard treatment

INTERVENTIONS:
Other: standard treatment — The control group will be provided with the necessary approaches for diabetic foot ulcer care and diaphragmatic breathing exercises.
  Other Names: control
  Arms: control group
Other: aerobic exercise — The aerobic exercise group will be provided with the necessary approaches for diabetic foot ulcer care and in addition to diaphragmatic breathing exercises, they will be provided with aerobic exercise twice a week with a physiotherapist.
  Arms: aerobic exercise group
Other: exercise protocol — The protocol exercise group will be provided with the necessary approaches for diabetic foot ulcer care and exercises suitable for the physical condition of the wound and the patient, in addition to diaphragmatic breathing exercises. This group will also work with a physiotherapist twice a week.
  Arms: exercise protocol group

SUMMARY:
Exercise studies with patients with diabetic foot ulcers are very few. In this disease group, since it is considered dangerous to put a load on the foot, a barrier has been placed between the patients and the exercise. With the study investigators plan to do, investigators will try to exercise in these patients in a controlled manner. Among the patients divided into 3 groups, the 1st group will apply the control group, the 2nd group will perform aerobic exercise, and the 3rd group will apply the exercises investigators have determined as the protocol group. 12 weeks, 2 sessions a week will be exercised with the help of a physiotherapist. Patients will be evaluated at baseline, at the end of week 4, at the end of week 8, and at the end.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with Type II diabetes and having a foot ulcer
* Being in the 1st or 2nd category according to the Wagner classification
* Not to have a serious musculoskeletal, cardiac, neurological, etc. systemic disease that may interfere with the research.
* Not having any communication problems
* Having the same wound care procedure
* Not taking any other treatment that may have an effect on the wound.

Exclusion Criteria:

* Individuals with a diagnosed psychiatric illness,
* Individuals who have received any physiotherapy treatment in the last 3 months,
* Individuals with acute infection,
* Individuals with toe pressure < 40 mmHg
* Individuals with Charcot Foot and/or osteomyelitis
* Individuals with venous ulcer disease
* Individuals who are morbidly obese (BMI >40) according to body mass index
* Individuals with incurable proliperative retinopathy

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
ulcer area (mm²) | initial assessment- 4th week- 8th week- 12th week
  Calculation of ulcer area with image j program
ulcer depth (mm) | initial assessment - 12th week
  Ulcer depth measurement with sterile wound stick

SECONDARY OUTCOMES:
quality of life score | initial assessment - 12th week
  Investigation of patients' quality of life with Ferrans&Powers quality of life index
sleep quality score | initial assessment - 12th week
  investigating the sleep quality of patients with the Pittsburgh sleep quality index

OTHER OUTCOMES:
kinesiophobia score | initial assessment - 12th week
  Investigation of patients' fear of movement with TAMPA

CONTACTS AND LOCATIONS:
Locations (1):
- Harran Unıversıty, Sanliurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR